CLINICAL TRIAL: NCT06414460
Title: A Phase 1, Open-Label, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Preliminary Efficacy of ISM3412 in Participants With Locally Advanced/Metastatic Solid Tumors
Brief Title: Study of ISM3412 in Participants With Locally Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISM3412-101
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced/Metastatic Solid Tumors
Keywords: Methionine adenosyltransferase 2A (MAT2A); homozygous MTAP deletion; MAT2A inhibitor; ISM3412

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Dose Escalation (Experimental): Patients will receive ISM3412 once daily in sequential cohorts of increasing doses.
  Interventions: Drug: ISM3412
- Part 2 Dose Selection Optimization (Experimental): Participants will be randomized to receive one of the two selected dose levels of ISM3412 once daily determined by Study Review Committee.
  Interventions: Drug: ISM3412

INTERVENTIONS:
Drug: ISM3412 — ISM3412 will be administered orally once daily.

SUMMARY:
The study has consists of two parts, a dose escalation part (Part 1) and a dose selection optimization part (Part 2). The primary objectives of this study are to evaluate the safety and tolerability of ISM3412 in participants with locally advanced/metastatic solid tumors, and to determine the RP2D of ISM3412.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with age ≥18 years at the time of signing the informed consent.
2. Histologically confirmed unresectable locally advanced or metastatic solid tumors with confirmed homozygous MTAP deletion, who have disease progression after standard therapy, intolerable to standard therapy, or for whom no standard therapy exists.
3. Have measurable or evaluable lesions in Part 1 and at least one measurable target lesion in Part 2 as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
4. Participants must provide a documentary evidence of homozygous MTAP deletion; or provide archival formalin-fixed paraffin-embedded (FFPE) tumor tissue blocks or at least 15 FFPE tumor tissue slides, or perform tumor tissue biopsies for a confirmatory genetic test indicating homozygous MTAP deletion.
5. ECOG PS (Eastern Cooperative Oncology Group Performance Status) ≤1.
6. Life expectancy of ≥12 weeks as judged by the investigator.
7. Adequate organ function as determined by medical assessment.
8. Capable of providing signed ICF and complying with the requirements and restrictions listed in the ICF and in this study protocol.

Exclusion Criteria:

1. Prior treated with other MAT2A inhibitors and/or PRMT inhibitors.
2. Participation in other therapeutic clinical studies within 28 days or 5 half-lives (whichever is shorter) prior to first dose of study treatment.
3. Anti-tumor therapy (chemotherapy, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, or other anti-tumor therapy, except for hormones for hypothyroidism or estrogen replacement therapy, anti-estrogen analogues, agonists required to suppress serum testosterone levels) within 28 days or 5 half-lives, whichever is shorter prior to first dose of study treatment.
4. Toxicities of prior therapy have not resolved to Grade ≤1 or to baseline (as evaluated by NCI CTCAE version 5.0)
5. History of another primary tumor that has been diagnosed or required therapy within the past 3 years.
6. Previous history of, or presence of Gilbert's syndrome.
7. Previous history of myelodysplastic syndrome.
8. Prior solid organ or hematopoietic stem cell transplant.
9. Known active central nervous system (CNS) primary tumor or untreated CNS metastases.
10. Have serious cardiovascular or cerebrovascular disease as per protocol.
11. Presence of uncontrolled systemic infection as per protocol.
12. Unwillingness or unable to comply with the requirements of oral drug administration, or presence of a gastro-intestinal condition.

Other protocol inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) events | 31 days
  To evaluate the safety and tolerability of ISM3412.
Incidence and severity of adverse events (AEs) | Approximately 30 months
  To evaluate the safety and tolerability of ISM3412.
Recommended phase 2 dose (RP2D) | Approximately 30 months
  To determine the RP2D of ISM3412.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Approximately 30 months
  To assess PK of ISM3412 in plasma following a single and multiple doses of ISM3412
Time of maximum observed concentration (Tmax) | Approximately 30 months
  To assess PK of ISM3412 in plasma following a single and multiple doses of ISM3412
Area under the concentration-time curve (AUC) | Approximately 30 months
  To assess PK of ISM3412 in plasma following a single and multiple doses of ISM3412
Terminal half-life (t1/2) | Approximately 30 months
  To assess PK of ISM3412 in plasma following a single and multiple doses of ISM3412
Objective response rate (ORR) | Approximately 30 months
  To evaluate the preliminary efficacy of ISM3412 in participants with locally advanced/metastatic solid tumors.
Best objective response (BOR) | Approximately 30 months
  To evaluate the preliminary efficacy of ISM3412 in participants with locally advanced/metastatic solid tumors.
Duration of response (DoR) | Approximately 30 months
  To evaluate the preliminary efficacy of ISM3412 in participants with locally advanced/metastatic solid tumors.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (5):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Smilow Cancer Hospital at Yale New Haven Breast Center, New Haven, Connecticut
  - Community Cancer Center North, Indianapolis, Indiana
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen university cancer center, Guangzhou, Guangdong
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Shanghai Gobroad Cancer Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No